CLINICAL TRIAL: NCT01318395
Title: Randomized, Double Blind, Active-controlled, Parallel Study to Analyse Effects of the Combination of Aliskiren and Valsartan on the Vascular Structure and Function of Retinal Vessels
Brief Title: Aliskiren on Retinal Vasculature Treatment Study
Acronym: ARTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100ADE07T
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Active Comparator)
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — orally 150 mg/d for 1 week, then orally 300 mg/d for 7 weeks
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Placebo — orally once per day
  Arms: Placebo

SUMMARY:
Hypertension affects approximately one fourth of the world population and therefore contributes substantially to the worldwide burden of cardiovascular (CV) disease and end-organ damage.

Changes in small artery structure characterized by an increased wall-to-lumen ratio (WLR) are characteristic feature of target organ damage in hypertension. Of clinical importance, structural arteries of small subcutaneous arteries have been shown to be of prognostic significance, with adverse prognosis in subjects with higher WLR. However, the assessment of arteriolar structure from biopsies of subcutaneous tissue is invasive and impractical in clinical practice. A new approach focuses on retinal arteriolar structural parameters by using scanning laser Doppler flowmetry (SLDF) with automatic full-field perfusion imaging analyses (9). This approach allows the non-invasive assessment of both the outer diameter (OD) and inner diameter (ID) of retinal arterioles in vivo and, thus, analyses vascular remodeling of retinal arterioles by calculating WLR = (OD - ID) / ID).

A crucial role in the efforts of prevention of end-organ damage plays the renin angiotensin system (RAS). The increased mechanical strain on the vasculature at a higher BP can cause injury to the endothelial wall. Activation of the RAS increases BP and stimulates a local inflammatory response to repair the injury. Long-term or repeated response to injury leads to endothelial dysfunction and microvascular damage, and hence end-organ damage.

Combining RAS inhibitors may provide greater end-organ protection than use of either class alone. However, ONTARGET has failed to show superiority of the dual RAS blockade (ACE-I and ARB) in patients at high cardiovascular risk. The combination of ARBs and direct renin inhibitors (DRIs) emerged as the only available, valid and innovative option for blocking the RAS at two different sites (sequential blockade). Indeed, AVOID study and ALLAY study demonstrated that the DRI aliskiren has additional and to some extent blood pressure independent effects on albuminuria and left ventricular hypertrophy, both signs of subclinical organ damage in hypertension, respectively.

However, no data are available with respect to the effects of ARBs and DRIs on vascular properties in the short and long term To close this gab we focus in this study on vascular structural and functional changes since vascular adaptation to high blood pressure occurs in the early phase of hypertensive disease.

DETAILED DESCRIPTION:
Hypertension affects approximately one fourth of the world population and therefore contributes substantially to the worldwide burden of cardiovascular (CV) disease and end-organ damage (1). Therefore, the goal of antihypertensive therapy is to provide effective long-term lowering of elevated blood pressure (BP) and prevention of hypertensive end-organ-damage and mortality (2).

Changes in small artery structure characterized by an increased wall-to-lumen ratio (WLR) are characteristic feature of target organ damage in hypertension. (3; 4). A clinical study examining small arteries obtained from gluteal biopsies of patients with hypertension revealed that an increased WLR of subcutaneous small arteries is one of the first manifestations of target organ damage in hypertension that occur before proteinuria and cardiac hypertrophy (5). Of clinical importance, structural arteries of small subcutaneous arteries have been shown to be of prognostic significance, with adverse prognosis in subjects with higher WLR (6-8). However, the assessment of arteriolar structure from biopsies of subcutaneous tissue is invasive and impractical in clinical practice. A new approach focuses on retinal arteriolar structural parameters by using scanning laser Doppler flowmetry (SLDF) with automatic full-field perfusion imaging analyses (9). This approach allows the non-invasive assessment of both the outer diameter and inner diameter of retinal arterioles in vivo and, thus, analyses vascular remodeling of retinal arterioles by calculating WLR = (outer diameter - inner diameter) / inner diameter) (10).

In a previous study, we could demonstrate that treated hypertensive patients with poor BP control have a greater WLR of retinal arterioles than those with good blood pressure control. Interestingly, in this cohort we did not find a significant relation between BP and WLR of retinal arterioles using correlation analyses. We have concluded that this lack of a relation might well be the result of the effects of some antihypertensive drugs to beneficially influence vascular structure (9). Subsequently, we analyzed WLR of retinal arterioles in a cohort of never-treated patients with essential hypertension and normotensive controls. In this cohort, both systolic BP and diastolic BP were significantly related to WLR of retinal arterioles independent of traditional CV risk factors and other confounders, e.g. subclinical inflammation, endothelial dysfunction and dietary salt intake. Moreover, in this cohort, the WLR of retinal arterioles was greater in hypertensive than in normotensive subjects (11).

A crucial role in the efforts of prevention of end-organ damage plays the renin angiotensin system (RAS) due its dual role on salt and water homeostasis (blood pressure) and the vascular response to injury. The increased mechanical strain on the vasculature at a higher BP can cause injury to the endothelial wall. Activation of the RAS increases BP and stimulates a local inflammatory response to repair the injury. Long-term or repeated response to injury leads to endothelial dysfunction and microvascular damage (12), and hence end-organ damage. Therefore increasing evidence is not suppressing, that antihypertensive medications which inhibit the RAS may provide incremental end-organ protection.

Recently, we have shown that hypertensive patients have an impaired vasodilatory response of retinal arterioles to Flickerlight test - which improves after treatment with Angiotensin Receptor Blockers (ARBs) - and have a reduced nitric oxide (NO) activity in the retinal circulation, that is normalized after treatment with ARBs (13; 14). Likewise, in a previous study analyzing the arterial resistance vessels also in the systemic circulation we found that in contrast to diuretics and placebo, valsartan improved endothelial function and vascular properties (estimated by pulse wave anlalysis) (15; 16).

Combining RAS inhibitors may provide greater end-organ protection than use of either class alone. However, the Ongoing Telmisartan Alone and in Combination with Ramipril Global Endpoint Trial (ONTARGET) has failed to show superiority of the dual RAS blockade (Angiotensin converting enzyme inhibitor and ARB) in patients at high cardiovascular risk (17). The combination of ARBs and direct renin inhibitors (DRIs) emerged as the only available, valid and innovative option for blocking the RAS at two different sites (sequential blockade). Indeed, the Aliskiren in the Evaluation of Proteinuria in Diabetes (AVOID) study (18) and the Aliskiren in Left Ventricular Hypertrophy (ALLAY) study (19) demonstrated that the DRI aliskiren has additional and to some extent blood pressure independent effects on albuminuria and left ventricular hypertrophy, both signs of subclinical organ damage in hypertension, respectively (20).

However, no data are available with respect to the effects of ARBs and DRIs on vascular properties in the short and long term To close this gab we focus in this study on vascular structural and functional changes since vascular adaptation to high blood pressure occurs in the early phase of hypertensive disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years (females of child bearing potential must be using adequate contraceptive precautions)
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at enrolment visit
* Patients with mild to moderate uncomplicated essential hypertension with a trough mean sitting DBP ≥ 90 mmHg and/or SBP ≥ 140 mmHg or pretreated arterial hypertension
* Written informed consent
* Agreement to attend all study visits as planned in the protocol
* Agreement to perform routinely self home blood pressure measurements as well as keep a blood pressure diary throughout the study and to inform the investigator if BP exceeds cutt off criteria given in the ICF

Exclusion Criteria:

* In the investigator's opinion the patient can not be withdrawn from their current antihypertensive medication
* Secondary hypertension (e.g. patients with hyperaldosteronism, pheochromocytoma, renal artery stenosis, renal parenchymal disease, coarctation of the aorta, Cushing's disease syndrome)
* Severe essential hypertension (systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg) or treatment resistant hypertension (3 antihypertensive drugs and still SBP ≥ 140mmHg and/or DBP ≥ 90mmHg)
* History of hypertensive encephalopathy or intracerebral hemorrhage
* Diabetes mellitus Type 1 or Type 2
* History of epilepsia (no retinal exam possible)
* Eye cataract (no retinal exam possible)
* History of the following within the last six months: myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, heart failure
* Presence of significant renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, immunological, haematological or oncological, neurological and psychiatric diseases or dysfunction
* Impaired renal function as shown by estimated GFR (abbreviated MDRD formula) < 45 ml/min/1.73 m2
* Impaired hepatic function as shown by transaminases higher than three times the upper normal limit
* Known allergy or a known intolerance to any ARB or Aliskiren
* Females who are pregnant or lactating or who are not on an adequate contraception (Pearl-Index ≥ 1 %)
* Use of any investigational drug within 28 days before study entry
* Patients previously enrolled into the study
* History of drug, medication abuse.
* Serious disorders which may limit the ability to evaluate the efficacy or safety of the test drug(s), including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, immunological, haematological or oncological, neurological and psychiatric diseases
* Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Subject unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up visits and unlikelihood of completing the study
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To investigate the combined effect of aliskiren and valsartan on vascular structure, assessed by wall to lumen ratio of retinal arterioles, in hypertensive patients. | After 8 weeks of treatment with aliskiren versus placebo
  WLR = (outer diameter - inner diameter) / inner diameter) of retinal arterioles

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (2):
- Germany (2):
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen
  - Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Nuremberg

REFERENCES:
- [Result] Jumar A, Ott C, Kistner I, Friedrich S, Schmidt S, Harazny JM, Schmieder RE. Effect of aliskiren on vascular remodelling in small retinal circulation. J Hypertens. 2015 Dec;33(12):2491-9. doi: 10.1097/HJH.0000000000000735. PMID 26398851
- [Derived] Bosch A, Schmid A, Ott C, Kannenkeril D, Karg MV, Ditting T, Veelken R, Uder M, Schmieder RE. Copeptin Levels in Patients With Treatment-Resistant Hypertension Before and 6 Months After Renal Denervation. Am J Hypertens. 2020 Feb 22;33(2):182-189. doi: 10.1093/ajh/hpz155. PMID 31555795
- [Derived] Bosch AJ, Harazny JM, Kistner I, Friedrich S, Wojtkiewicz J, Schmieder RE. Retinal capillary rarefaction in patients with untreated mild-moderate hypertension. BMC Cardiovasc Disord. 2017 Dec 21;17(1):300. doi: 10.1186/s12872-017-0732-x. PMID 29268712